CLINICAL TRIAL: NCT03189550
Title: Enhanced Recovery After Surgery in Colorectal Surgery: A Large-Scale Quality Improvement Project
Acronym: ERAS
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Matthew McEvoy, Associate Professor of Anesthesiology, Vanderbilt University Medical Center
Other Study IDs: 140558
Record Dates: First submitted 2017-03-25; First posted 2017-06-16 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Surgery; Quality Improvement; Perioperative Care; ERAS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Historical control: Patients who underwent colorectal surgery with standard perioperative care starting from June 2014 and progressing backward in time.
  Interventions: Procedure: Standard perioperative care
- ERAS without SOC noninvasive hemodynamic monitoring: Patients who underwent colorectal surgery after implementation of standard of care (SOC) ERAS perioperative care from July 2014 to February 2015
  Interventions: Procedure: ERAS perioperative care; Procedure: Standard perioperative care
- ERAS with SOC noninvasive hemodynamic monitoring: Patients who underwent colorectal surgery after implementation of standard of care ERAS perioperative care with standard of care noninvasive hemodynamic monitoring (with the ClearSight System, Edwards Lifesciences) after February 2015
  Interventions: Procedure: ERAS perioperative care; Procedure: Standard perioperative care; Procedure: Noninvasive hemodynamic monitoring

INTERVENTIONS:
Procedure: ERAS perioperative care — Standard of care implementation of multi-modal evidence-based care pathway, including standardized preoperative preparation (medical and diet), perioperative goal-directed fluid therapy, multi-modal perioperative pain management, postoperative nausea and vomiting prevention, surgical care and bowel isolation, and surgical site infection prevention
  Groups: ERAS with SOC noninvasive hemodynamic monitoring; ERAS without SOC noninvasive hemodynamic monitoring
Procedure: Standard perioperative care — Standard perioperative care prior to implementation of ERAS care pathway
Procedure: Noninvasive hemodynamic monitoring — Standard of care perioperative noninvasive hemodynamic monitoring with the ClearSight System (Edwards LifeSciences)
  Groups: ERAS with SOC noninvasive hemodynamic monitoring

SUMMARY:
Multimodal perioperative care pathways have evolved into enhanced recovery after surgery (ERAS). ERAS pathways improve the quality of patient care, reduce morbidity, and shorten length of stay. This project will test the hypothesis that implementation of a multi-modal ERAS perioperative care protocol in colorectal surgical patients will result in significantly reduced perioperative morbidity and mortality.

DETAILED DESCRIPTION:
Multimodal perioperative care pathways have evolved into enhanced recovery after surgery (ERAS). ERAS pathways improve the quality of patient care, reduce morbidity, and shorten length of stay. This large quality improvement project will compare outcomes after standard perioperative practice with those after the implementation of a multi-modal evidence based care pathway, including standardized preoperative preparation, perioperative goal-directed fluid therapy (GFDT), multi-modal perioperative pain management, post operative nausea and vomiting prevention, surgical care and bowel isolation, and surgical site infection prevention. This project will test the hypothesis that implementation of a multi-modal ERAS perioperative care protocol in colorectal surgical patients will result in significantly reduced perioperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent colorectal surgery at Vanderbilt University Medical Center and whose data is stored in the perioperative data warehouse.

Exclusion Criteria:

* Age <18 years
* Weight <40 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent colorectal surgery at Vanderbilt University Medical Center
Sampling Method: Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical site infection | Up to 30 days postoperative

SECONDARY OUTCOMES:
ICU length of stay | Up to 30 days postoperative
Time on ventilator | Up to 30 days postoperative
Post operative pain assessment using 11-point Numeric Pain Rating Scale (NRS) | Up to 30 days postoperative
  Post operative pain assessed using NRS when 0 is no nausea and 10 is worst pain.
Post operative anti emetic consumption | Up to 30 days postoperative
Occurrence of postoperative complications | Up to 30 days postoperative
Analgesia consumption | Up to 30 days postoperative
  Total opioid and non-opioid medication use
Cardiac Index | 1 day
  Using time traces for cardiac index during the perioperative period, the time in range of pre-defined parameters will be measured.
Stroke volume | 1 day
  Using time traces for stroke volume during the perioperative period, the time in range of pre-defined parameters will be measured.
Systemic vascular resistance | 1 day
  Using time traces for systemic vascular resistance during the perioperative period, the time in range of pre-defined parameters will be measured.
Heart rate | 1 day
  Using time traces for heart rate during the perioperative period, the time in range of pre-defined parameters will be measured.
Hospital Length of stay (days) | Up to 30 days post operative

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D McEvoy, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McEvoy MD, Wanderer JP, Shi Y, Ramanujan KS, Geiger TM, Shotwell MS, Shaw AD, Hawkins AT, Martin BJ, Mythen MG, Sandberg WS. The effect of adding goal-directed hemodynamic management for elective patients in an established enhanced recovery program for colorectal surgery: results of quasi-experimental pragmatic trial. Perioper Med (Lond). 2020 Nov 23;9(1):35. doi: 10.1186/s13741-020-00163-3. PMID 33292514